CLINICAL TRIAL: NCT04308629
Title: Cortical Enhancement of Posture, Movement Planning, and Execution of Upright Reaching Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Sandy McCombe Waller, Principle Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00064894
Record Dates: First submitted 2020-03-03; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-02

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: StartReact response; transcranial direct current stimulation; Postural control
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS over PMAs (Experimental): One session of transcranial direct current stimulation (tDCS) over premotor areas (PMAs)
  Interventions: Other: Transcranial direct current stimulation
- tDCS over M1 (Active Comparator): One session of transcranial direct current stimulation (tDCS) over primary motor area (M1)
  Interventions: Other: Transcranial direct current stimulation

INTERVENTIONS:
Other: Transcranial direct current stimulation

SUMMARY:
Stroke is the leading cause of disability and diminished quality of living that frequently includes impairments of postural control and upper extremity (UE) function. The interaction of posture and UE coupling in terms of movement planning, initiation, and execution is not well understood. StartReact responses triggered by a loud acoustic stimulus (LAS) during the planning and preparation of goal intended actions has been used to probe the state of brainstem neuronal excitability related to posture and movement sequencing. The purpose of this study is to examine posture and goal-directed movement planning and execution using startReact responses and to evaluate posture and UE movement sequence during reaching while standing in individuals with chronic hemiparesis and healthy controls. Secondly, the investigators will determine the modulatory role of the cortical premotor areas (PMAs) in startReact responses in healthy controls and in persons with stroke by using transcranial direct current stimulation (tDCS) to up- or down-regulate PMAs excitability.

ELIGIBILITY:
Inclusion Criteria for stroke:

* Unilateral cortical or white matter subcortical stroke
* Age 40 yrs and older
* ≥ 6 months post ischemic stroke or ≥ 12 months post hemorrhagic stroke
* Residual arm hemiparesis as indicated by Fugl-Meyer Upper Extremity score between 20-65
* Having the ability to perform reaching movements with the paretic arm in standing without an assistive device.

Exclusion Criteria for stroke:

* Stroke involving bilateral hemisphere, brainstem or cerebellum
* Any medical condition precluding participation in testing
* Other health conditions affecting balance and upper extremity movement function beyond the effects of stroke.

Inclusion Criteria for healthy controls:

* Age-matched to the stroke subjects
* Without a history of stroke or any known neurological conditions
* Having the cognitive ability to follow two-step commands and give informed consent

Exclusion Criteria for healthy controls:

* Any medical condition precluding participation in testing
* Other health conditions affecting balance and upper extremity movement function beyond the effects of stroke.

Participants were also excluded if they did not meet the TMS safety criterion including having implantable medical devices, history of seizures, taking medications to reduce anxiety, sedatives, and seizure, and pregnancy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Change in startReact response | Immediately after the intervention (one session tDCS)
  The incidence of StartReact response following an loud acoustic stimulus
Change in the lag between anticipatory postural adjustments and reach onset | Immediately after the intervention (one session tDCS)
  The temporal lag between anticipatory postural adjustments (APA) onset and reach onset (unit: seconds)

SECONDARY OUTCOMES:
Change in the reach onset (unit: seconds) | Immediately after the intervention (one session tDCS)
  The onset of the anterior wrist joint center movement with a threshold of 5% peak velocity
Change in the APA onset (unit: seconds) | Immediately after the intervention (one session tDCS)
  The onset of the posterior center of pressure displacement with a threshold of 5% peak velocity
Change in the amount of trunk flexion (unit: radians) | Immediately after the intervention(one session tDCS)
  The angular displacement of the line joining the reaching shoulder and the hip joint center on the same side in the sagittal plane at maximum reach normalized by reach distance
Change in the amount of trunk rotation (unit: radians) | Immediately after the intervention (one session tDCS)
  The angular displacement of the line connecting both shoulders in the horizontal plane in the direction of the reach at maximum reach normalized by reach distance
Change in the amount of pelvic rotation (unit: radians) | Immediately after the intervention (one session tDCS)
  The angular displacement of the line connecting both hip joint centers in the horizontal plane in the direction of the reach at maximum reach normalized by reach distance
Change in the amount of trunk-pelvic rotation difference (unit: radians) | Immediately after the intervention (one session tDCS)
  The difference between trunk and pelvic angular displacement at maximum reach normalized by reach distance

REFERENCES:
- [Derived] Yang CL, Gad A, Creath RA, Magder L, Rogers MW, Waller SM. Effects of transcranial direct current stimulation (tDCS) on posture, movement planning, and execution during standing voluntary reach following stroke. J Neuroeng Rehabil. 2021 Jan 7;18(1):5. doi: 10.1186/s12984-020-00799-8. PMID 33413441